CLINICAL TRIAL: NCT00470717
Title: Early Feeding and Wellness Among Late Preterm Infants Born at MacDonald Women's Hospital: A Feasibility Study for a Breastfeeding Intervention
Brief Title: Feeding and Wellness Among Late Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Lydia Furman, Physician, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LF-UH-1001
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Late Preterm Infant
Keywords: late preterm infant; breastfeeding; formula feeding; rehospitalization; telephone
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phone calling (Other): Weekly telephone call. There are not two arms to the study. The primary intervention is phone calling weekly to assess ability to complete phone call and obtain feeding data.
  Interventions: Procedure: Weekly telephone call

INTERVENTIONS:
Procedure: Weekly telephone call — Details of feeding and health/sickness will be obtained

SUMMARY:
1. The first aim of this proposal is to pilot the feasibility of weekly phone monitoring of infant feeding and illness patterns in a socio-economically and racially diverse population. Specifically, the investigators aim to estimate the rate of group loss to follow up from birth to 13 weeks (3 months) of age with weekly phone interview of mothers of late preterm (LPT, gestational age 34 0/7- 36 6/7 weeks gestation) infants.
2. The second aim is to describe breastfeeding and formula feeding practices, and rates of illness and post-discharge hospital care utilization, through age 13 weeks (3 months) among late preterm infants born at MacDonald Women's Hospital. The investigators estimate that the rate of exclusive breastfeeding among LPT infants at 3 months of age is less than the documented rate of 37% for all infants in Cuyahoga County.

DETAILED DESCRIPTION:
Late preterm infants (LPT, gestational age 34 0/7 - 36 6/7 weeks) are the largest proportion of all preterm (less than 37 weeks gestation) infants. Recent evidence finds an increased risk of early post-discharge morbidity and re-hospitalization among LPT as compared to full term infants, which is linked to breastfeeding, specifically to early lactation failure and decreased breast milk intake. Accurate and inexpensive methods to collect data on rates of breastfeeding and early morbidity among LPT infants are critical to design, implementation and monitoring of effective interventions. This pilot study evaluates the feasibility of weekly phone calling in a racially and socioeconomically diverse population of mothers of LPT infants.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of singleton LPT (late preterm, gestational age 34 0/7- 36 6/7 completed weeks) infants

Exclusion Criteria:

* Exclusion criteria for mothers include positive maternal drug screen for drug of abuse
* Age < 18 years, or per caregiver discretion mother is not appropriate for study.
* Exclusion criteria for infants include custody under contention, positive screen for maternal drugs of abuse, or major congenital anomaly or congenital infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia M Furman, M.D., Principal Investigator — Case Western Reserve University School of Medicine
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 84 inborn LPT infants admitted, 68 (81%) were eligible of whom 39 (57%) agreed to participate, 27 declined and 2 were missed due to brief hospital stays. Sixteen were ineligible: teen mother (7), major congenital malformation (3), positive maternal toxicology screen (2), custody uncertain/other reason (4).
Pre-assignment Details: One infant was withdrawn from the study due to an unexpectedly long hospital stay (>13 weeks), yielding a total of 38 study infants.
Units Other Than Participants: phone call attempts
Groups:
- Phone Calling: Weekly telephone call. There are not two arms to the study. The primary intervention was phone calling weekly to assess ability to complete phone call and obtain feeding data.
  Weekly telephone call: Details of feeding and health/sickness were obtained
Period: Overall Study
Arm/Group | Phone Calling
Started (Milestone is beginning enrollment) | 38; 1976 phone call attempts (Each participant could be called up to 4 times weekly for 13 weeks (38x4x13))
Completed (End of calling attempts) | 38; 813 phone call attempts
Not Completed | 0; 1163 phone call attempts

BASELINE CHARACTERISTICS:
Arm/Group | Phone Calling
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants] — mean age of 26.8 years (SD = 6.1)
  Participants
    <=18 years | 0
    Between 18 and 65 years | 38
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Phone Call Completion Rate
Description: Phone call Completion is defined as the phone call was answered by the participant and information was obtained on the survey measures. Phone call completion rate is the number of calls completed over the study period.
Time Frame: Time frame: 13 weeks (3 months)
Measure: Number; unit: calls
Units Other Than Participants: phone call
Arm/Group | Phone Calling
Number analyzed (Participants) | 38
Number analyzed (phone call) | 494
calls
  Reached with one call over 13 weeks | 194
  Reached with 2 calls over 13 weeks | 102
  Reached with 3 or 4 calls over 13 weeks | 59
  Could not be reached with 4 calls over 13 weeks | 52
  Missing | 87

ADVERSE EVENTS:
Arm/Group | Phone Calling
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phone Calling (N=38)
loss of confidentiality (General disorders) | 0 (0) — The primary adverse event for this study would be loss of confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes